CLINICAL TRIAL: NCT07164963
Title: Upper Cervical Translatoric Mobilization Versus Sub Occipital Muscle Energy Technique in Patients With Mechanical Neck Pain and Forward Head Posture
Brief Title: Upper Cervical Mobilization vs. Sub-Occipital MET for Neck Pain and FHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, reda abd elrazik, Associate Professor, Department of Physical Therapy, Faculty of Physical Therapy, Benha University, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT.BU.EC.22
Record Dates: First submitted 2025-08-31; First posted 2025-09-10 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Mechanical Neck Pain; Forward Head Posture
Keywords: Mechanical Neck Pain; Forward Head Posture; Upper Cervical Mobilization; Muscle Energy Technique; Craniovertebral Angle; Neck Disability Index

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Upper Cervical Translatoric Mobilization (Experimental): Participants will receive Upper Cervical Translatoric Mobilization (UC-TSM) applied to the upper cervical spine (C0-C2), in addition to conventional physical therapy (hot pack and Kendall exercises), three times per week for 4 weeks.
  Interventions: Other: upper cervical translatoric mobilisation
- Sub-Occipital Muscle Energy Technique (Experimental): Participants will receive Sub-Occipital Muscle Energy Technique (MET) targeting the sub-occipital muscles, in addition to conventional physical therapy (hot pack and Kendall exercises), three times per week for 4 weeks.
  Interventions: Other: sub occipital muscle energy technique
- traditional physical therapy (Active Comparator): Participants will receive conventional physical therapy only, including application of a hot pack for 15 minutes followed by Kendall exercises for postural correction, three times per week for 4 weeks.
  Interventions: Other: traditional physical therapy

INTERVENTIONS:
Other: upper cervical translatoric mobilisation — (UC-TSM) is defined as a system of manual techniques using straight-line forces delivered in a parallel or perpendicular direction to an individual vertebral joint or motion segment there is also increasing in body of evidence supporting the its clinical effectiveness and safety in the management of patients with cervical impairments.
  Arms: Upper Cervical Translatoric Mobilization
Other: sub occipital muscle energy technique — Muscle Energy Technique (MET) is another form of a gentle manual therapy intervention that primarily targets the soft tissues, though it also contributes significantly to joint mobilization. It has been reported that, adding MET to exercise program resulted in better improvement in CVA and FHP than exercise group only
  Arms: Sub-Occipital Muscle Energy Technique
Other: traditional physical therapy — hot pack and kendel exercise
  Arms: traditional physical therapy

SUMMARY:
forty-five patients with MNP and FHP age from 25-40 years will be randomly assigned into three groups: Group A (study): 15patients will receive (upper cervical translatoric mobilization) and traditional physical therapy, Group B (study): 15patients received sub occipital muscle energy technique and traditional physical therapy, and Group C (control): 15 patients will receive the traditional physical therapy treatment only . Interventions will be conducted three times a week for four weeks. Craniovertebral angle (CVA) using Photographic Posture Analysis Method (surgimap software), pain intensity using viual analogue scale (VAS), Cervical ROM using CROM device, and neck functional ability using Neck Disability Index (NDI) will be assessed for all participants before and after the treatment program.

DETAILED DESCRIPTION:
This randomized controlled trial aims to compare the efficacy of Upper Cervical Translatoric Mobilization (UC-TSM) and Sub-Occipital Muscle Energy Technique (MET) in patients with Mechanical Neck Pain (MNP) and Forward Head Posture (FHP). Forty-five participants will be randomly assigned to one of three groups: Group A (UC-TSM + conventional physical therapy), Group B (Sub-Occipital MET + conventional physical therapy), and Group C (conventional physical therapy only). Interventions will be administered three times per week for four weeks. Outcomes include pain intensity (VAS), neck disability (NDI), cervical range of motion (CROM), and craniovertebral angle (CVA) assessed via photographic analysis (Surgimap). The study will be conducted at Benha University.

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 20-60 Years
* suffering from M echanical neck pain with Craniovertebral angle ; < 53
* their NDI ranging from 30-48% [9]. Patients were excluded from the study if they have injury or trauma to cervical region, spinal surgery, cervical canal stenosis, radicular pain and malignancy.

Exclusion Criteria:

* Patients were excluded from the study if they have injury or trauma to cervical region, spinal surgery, cervical canal stenosis, radicular pain and malignancy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2025-09-12 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for Pain Intensity | Baseline and after 4 weeks of treatment
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a 10-cm line where 0 = "no pain" and 10 = "worst pain imaginable". A lower score indicates improvement.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) for Pain Intensity | Baseline and after 4 weeks of treatment
  Functional disability will be assessed using the Neck Disability Index (NDI), a 10-item questionnaire scored from 0 to 50, where higher scores indicate greater disability.
Craniovertebral Angle (CVA) via Photographic Posture Analysis | baseline and after 4 weeks
  The craniovertebral angle (CVA) will be measured using lateral-view photography and analyzed using Surgimap software. A higher CVA indicates improvement in forward head posture.

CONTACTS AND LOCATIONS:
Overall Officials: reda K. Abdelrazik, associate professor, Principal Investigator — Benha University
Locations (1):
- Faculty of Physical Therapy, Benha University, Cairo, Benha, Egypt

IPD SHARING:
Plan to Share IPD: No